CLINICAL TRIAL: NCT03509324
Title: Effectiveness and Determinants of Glucose Control, β-cell Function in Response to Short-term Intensive Insulin Pump Therapy in Different Duration of Type 2 Diabetes Mellitus.
Brief Title: Effectiveness of Glucose Control, β Cell Function in Response to Short-term Insulin Pump Therapy in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanbing Li, Director of Endocrinology Department, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMT20150410
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- duration of disease (Other): different duration of disease receive insulin LISPRO
  Interventions: Drug: Insulin LISPRO

INTERVENTIONS:
Drug: Insulin LISPRO — receive short-term insulin pump therapy by using insulin LISPRO, continue treatment for 7 more days when euglycemia achieved
  Other Names: humalog

SUMMARY:
The purpose of this study is to investigate and evaluate the significance of intravenous glucose tolerance test in assessment of β-cell function improvement after short course of intensive insulin therapy, trying to illustrate the relationship between fasting plasma glucose and acute insulin release under different stage of type 2 diabetes with poor glycemic control.

ELIGIBILITY:
Inclusion Criteria: different course of type 2 diabetes with poor glycemic control

-

Exclusion Criteria:

* acute complication or severe comorbidities

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
fasting plasma glucose after insulin therapy | 10 hour

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Li, MD,PhD, Principal Investigator — Ministry of Education
Locations (1):
- endocrinology department of the first affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China